CLINICAL TRIAL: NCT02851888
Title: Use of Regional Anesthesia in Hip Arthroscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Georgetown University (Other)
Collaborators: Union Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-0095
Record Dates: First submitted 2016-07-26; First posted 2016-08-02 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2017-11

CONDITIONS: Hip Injuries
MeSH Terms: conditions — Hip Injuries | interventions — Ropivacaine; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iliac Fascia Block (Ropivacaine) (Experimental): These patients will receive a preoperative iliac fascia block performed as a single shot in the standard fashion prior to hip arthroscopy with general anesthesia.
  Interventions: Drug: Ropivacaine; Procedure: General Anesthesia
- Control (Normal Saline Sham Injection) (Sham Comparator): These patients will receive a preoperative sham block of normal saline in the same fashion as a standard singl shot iliac fascia block prior to hip arthroscopy with general anesthesia.
  Interventions: Other: Normal Saline Sham Injection; Procedure: General Anesthesia

INTERVENTIONS:
Drug: Ropivacaine — Iliac fascia block was performed in the experimental group with a single shot of Ropavicaine.
  Other Names: Iliac Fascia Block
  Arms: Iliac Fascia Block (Ropivacaine)
Other: Normal Saline Sham Injection — Sham block using normal saline instead of iliac fascia block but otherwise employing the equivalent technique.
  Arms: Control (Normal Saline Sham Injection)
Procedure: General Anesthesia — Patients were induced and maintained in a fashion consistent with standard practices.

SUMMARY:
The purpose of this research is to determine differences in outcomes in patients who do, or do not, receive regional anesthesia (a fascia iliaca block) prior to undergoing hip arthroscopy with labral repair and/or debridement and osteoplasty for hip impingement

DETAILED DESCRIPTION:
Patients undergoing hip arthroscopy for hip impingement at the investigator's institution often have regional anesthesia (a nerve block) prior to the procedure to help prevent and/or reduce pain following the procedure. The investigators are interested in determining benefits as well as potential adverse effects of utilizing regional anesthesia in patients undergoing hip arthroscopy for impingement. To do so, they plan to enroll patients aged 18-50 undergoing hip arthroscopy, and randomize them to one of two groups with one group receiving regional anesthesia pre-operatively and the second control group, that does not. The surgical procedure and the post-operative management will be the same for both groups.

Regional anesthesia prior to orthopaedic procedures has been widely adopted in many fields of orthopaedics. While it is generally considered safe and an excellent adjuvant for pain control, there have been few studies exploring outcomes beyond pain control. In many centers, the use of regional anesthesia in hip arthroscopy is reserved for post-operative management of pain. There are multiple studies indicating that patients receiving regional anesthesia (a fascia iliaca or femoral nerve block) had significantly greater improvements in pain score and even an excellent alternative to routine narcotic medication in patients undergoing hip arthroscopy. Other orthopaedic procedures, such as knee arthroscopy, utilize similar techniques to achieve post-operative pain control through a femoral-sciatic nerve block.

There have also been studies looking at the utilization of regional anesthesia via lumbar plexus blocks with hip arthroscopy. One study found that patients undergoing hip arthroscopy with higher levels of preoperative psychological distress frequently utilized a lumbar plexus block to achieve adequate pain control. Other studies found that lumbar plexus blocks significantly improved pain while in the PACU. While serious complications of lumbar plexus block were rare, minor complications such as falls, persistent paresthesias, and unexpected admissions do occur. At our institution, we do not utilize lumbar plexus blocks for regional anesthesia in patients undergoing hip arthroscopy. Rather, our standard of care is to have an anesthesiologist perform a single shot fascia iliaca block using ropivicaine while the patient is in the pre-operative holding bay.

To the investigative team's knowledge, there are no studies comparing the difference in pain control, as well as the differences in narcotic requirements in PACU, duration of stay in PACU, reported falls, unplanned admissions and/or readmissions, Harris hip score and nerve pain/paresthesias/numbness in patients who have undergone hip arthroscopy with and without regional anesthesia. A better understanding of pain and functional outcomes following hip arthroscopy with and without regional anesthesia can help providers better assess circumstances when regional anesthesia can be beneficial or detrimental to a patient's post-operative course.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for arthroscopic labral repair with or without osteoplasty of the hip.
* 18 to 50 years old
* American Society of Anesthesiologists Physical Status (ASA PS) score of I or II.

Exclusion Criteria:

* Current or planned pregnancy
* History of neuropathic pain, chronic pain syndrome, or preoperative use of narcotic or neuropathic pain medicine
* Radiographic signs of osteoarthritis (> Tonis grade 1)
* Inability to attend follow up visits
* Documented allergy to local anesthetic

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-04 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Pain Medication Requirement in PACU | 24 hours post-operatively
  Measured in morphine equivalents

SECONDARY OUTCOMES:
Falls | 6 weeks
  patient reported
Readmissions | 6 weeks
  patient reported and through chart review
Neuropathic Pain | 2 weeks and 6 weeks
  Self Reported- Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS) questionnaires will be completed at both 2 and 6 week follow-up
Time to Physical Therapy | 6 weeks
  patient reported
Duration of PACU stay (mins) | 24 hours post-operatively
  time from PACU admission to discharge
Visual Analogue Pain Scores (VAS) | 24 hours post-operatively
  patient reported
Long Term Pain Control (daily VAS record) | 6 weeks
  Patients will complete a daily VAS questionnaire at home
Long Term Medication Requirements (daily log of medication usage in tablets of 5 mg oxycodone, morphine extended relief 15 mg, and/or indomethacin 75 mg) | 6 weeks
  Patients will complete a daily medication log at home
Modified Harris hip score | 6 weeks
  Questionnaire administered at 6 week follow up to evaluate functional outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Blake Bodendorfer, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No